CLINICAL TRIAL: NCT06252922
Title: A Pilot Study to Examine Metabolic Flexibility as a Mechanism for Diet- Induced Epigenetic Alterations in Male Gametes
Brief Title: Diet-Induced Changes in GEnetic Material
Acronym: DIG 'EM
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Emily W. Flanagan, MS, PhD, Postdoctoral Researcher, Pennington Biomedical Research Center
Other Study IDs: PBRC 2023-043
Record Dates: First submitted 2024-01-04; First posted 2024-02-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diet, Healthy; Body Weight; Metabolic Disturbance
Keywords: Healthy Weight; High-Fat Diet; Sperm DNA Methylation; Metabolic Flexibility; DNA Damage; Substrate Flux; Preconception
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot study in 10 men to test the hypothesis that perturbations in substrate flux and the circulating metabolic and pro-inflammatory milieus during a high-fat diet paradigm will modulate DNA methylation of genes in sperm associated with obesity and cardiometabolic dysfunction.

DETAILED DESCRIPTION:
The Paternal Origins of Health and Disease (POHaD) hypothesis was introduced to emphasize the need for research on paternal transmission of environmental exposures on offspring disease development. Paternal exposure to an obesogenic diet has been shown to imprint epigenetic predisposition to metabolic diseases which can be evident in offspring for up to 5 generations. In support, observational studies in men show that high-fat diets and diets high in processed foods significantly reduced the quantity and quality of sperm, including motility, morphology, and concentration, and DNA methylation of genes associated with obesity and cardiometabolic dysfunction. Yet, there are no experimental diet manipulation studies in males to understand the contribution of an acute obesogenic diet (i.e., high-fat) on DNA methylation of genes associated with obesity and cardiometabolic diseases in male gametes.

The research aims of this study are to: 1) measure DNA methylation of genes in semen in response to a healthy and high-fat diet, 2) examine metabolic flexibility in response to a healthy and high fat diet and its contribution to DNA methylation in semen, and 3) examine the metabolic and inflammatory milieu in response to a healthy and high fat diet and its contribution to DNA methylation in semen. To achieve these aims, we will conduct a cross-sectional, observational study in 10 healthy male participants 20-35 years of age using two diets (Healthy Diet: 27% Fat, 55% Carbohydrate, 15% Protein followed by a High-Fat Diet: 50% Fat, 35% Carbohydrate, 15% Protein).

ELIGIBILITY:
Inclusion Criteria:

* Male based on biological sex
* Age 20-35 years
* BMI between 18.5 and 24.9 kg/m2
* White/Caucasian
* Willing to consume pre-prepared meals
* Willing to wear an accelerometer and continuous glucose monitor (CGM)
* Willing to track diet intake
* Willing to stay 24 hours, including overnight in a research clinic
* Willing to provide blood and sperm samples
* Willing to consent to whole-genome sequencing of DNA

Exclusion Criteria:

* Unstable weight in the last 3 months (±5% weight loss or gain)
* Shift work or working in a factory setting
* Habitual smoking or use of tobacco products, including vaping, within the past 6 months.
* History of clinically diagnosed diabetes
* Hypertension (>140/90 mmHg measured at screening)
* Has undergone bariatric surgery
* History of cardiovascular disease, neurological disease, or other chronic diseases, including cancer
* History of human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
* Adherence to special or restrained diets (e.g., low-CHO, low-fat, or vegetarian/vegan diets) or food allergies associated with study foods.
* Currently engaging in >150 minutes moderate-intensity or >75 minutes of vigorous-intensity physical activity each week
* Drinking more than 14 servings of beer or alcohol per week
* Depressive (Score ≥10), anxiety (Score ≥8), and stress (Score≥15) symptomology (Score ≥16) from the 42-item Depression, Anxiety, Stress Scales (DASS)

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will enroll healthy men from the greater Baton Rouge area who meet the above eligibility criteria and are willing to participate in this research trial.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sperm DNA methylation | Baseline, Immediately after the healthy diet, Immediately after the high-fat diet
  Incidence of DNA methylation (whole genome/epigenome wide) of genes in sperm measured using bisulphate sequencing

SECONDARY OUTCOMES:
Sperm DNA Damage | Baseline, Immediately after the healthy diet, Immediately after the high-fat diet
  Comet Assay to determine DNA fragmentation in sperm.

OTHER OUTCOMES:
Metabolic Flexibility (indirect) | Immediately after the healthy diet, Immediately after the high-fat diet
  Change in respiratory quotient (RQ) from a fasted to a fed state using a metabolic chamber.
Metabolic Flexibility (direct) | Immediately after the healthy diet, Immediately after the high-fat diet
  Changes to circulating glucose from a fasted (0 minutes) to a fed state (240 minutes).
Continuous glucose monitoring | Immediately after the healthy diet, Immediately after the high-fat diet
  Mean Amplitude of Glycemic Excursions (MAGE) in response to healthy and high fat diets.
Insulin sensitivity | Immediately after the healthy diet, Immediately after the high-fat diet
  Mean 24hr glucose and total 24hr c-peptide excretion

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Official Study Landing Page — https://www.pbrc.edu/research-trials/view-all-current.aspx?studyid=402